CLINICAL TRIAL: NCT05108259
Title: A Phase 1, Double-blind, Randomized, Three-arm, Parallel Group Study to Compare the Pharmacokinetics and Safety of a Single Subcutaneous Dose of PBP1502, EU-Humira®, and US-Humira® in Healthy Male and Female Subjects.
Brief Title: To Compare the Pharmacokinetics and Safety of PBP1502 and Humira in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Prestige Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SOLOMON-I
Record Dates: First submitted 2021-10-01; First posted 2021-11-04 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers
Keywords: randomized; double-blind; phase 1
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PBP1502 (Experimental): Adalimumab single dose 40 mg (100 mg/mL) by SC injection via pre-filled syringe (PFS)
  Interventions: Drug: PBP1502
- EU-licensed Humira (Active Comparator): Adalimumab single dose 40 mg (100 mg/mL) by SC injection via PFS
  Interventions: Drug: EU-licensed Humira
- US-licensed Humira (Active Comparator): Adalimumab single dose 40 mg (100 mg/mL) by SC injection via PFS
  Interventions: Drug: US-licensed Humira

INTERVENTIONS:
Drug: PBP1502 — 40 mg/0.4 mL single SC injection via PFS
  Other Names: Adalimumab
  Arms: PBP1502
Drug: EU-licensed Humira — 40 mg/0.4 mL single SC injection via PFS
  Other Names: Adalimumab
  Arms: EU-licensed Humira
Drug: US-licensed Humira — 40 mg/0.4 mL single SC injection via PFS
  Other Names: Adalimumab
  Arms: US-licensed Humira

SUMMARY:
The main purpose of the study is to demonstrate pharmacokinetic (PK) equivalence of PBP1502 to the European (EU) and American (US) Humira reference products, following a single subcutaneous (SC) dose of 40 mg in healthy volunteers.

DETAILED DESCRIPTION:
This is a single centre, randomized, double-blind, three-arm, parallel group, single-dose, active comparator study, where a total of 324 healthy male and female adult volunteers - between the age of 18 and 55 years, both inclusive - will be dosed; 108 subjects per treatment group, randomly assigned to one of the 3 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects, between the age of 18 and 55 years, both inclusive (healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and heart rate measurement, 12-lead ECG, and clinical laboratory tests prior to administration of the study drug).
2. Subject is informed and able to understand the full nature and purpose of the study, including possible risks and side effects, and is given ample time and opportunity to read and understand this information. Subject has the ability and agrees to cooperate with the Investigator and must sign and date the written informed consent prior to performing any of the screening procedures.
3. BMI between 18.0 and 32.0 kg/m2, both inclusive.
4. Subject and their partner of childbearing potential must agree to use a highly effective method of contraception throughout the study and for 5 months after the administration of assigned treatment. A man is of childbearing potential if, in the opinion of the Investigator, he is sexually active. Male and female subjects and their partners who have been surgically sterilised for less than 24 weeks prior to the date of informed consent must agree to use any medically acceptable methods of contraception. Menopausal females must have experienced their last period more than 1 year prior to the date of informed consent to be classified as not of childbearing potential

Exclusion Criteria:

1. Subject has a medical history and/or condition including one or more of the following disease(s):

   * History and/or current presence of clinically significant atopy (e.g., allergic asthma, eczematous dermatitis), known or suspected clinically relevant hypersensitivity or allergic reactions to any of the excipients of study drug, other murine and human proteins, or Ig products.
   * Known infection with hepatitis B (active or carrier of hepatitis B), hepatitis C, or human immunodeficiency virus (HIV). However, a subject with history of hepatitis B virus is allowed if resolved.
   * History of invasive systemic fungal infections (including histoplasmosis, coccidioidomycosis, candidiasis, aspergillosis, blastomycosis, and pneumocystosis, etc.) or other opportunistic infections judged by the Investigator, including local fungal infections or a history of herpes zoster.
   * History of and/or current cardiac (including New York Heart Association class III/IV heart failure), gastrointestinal, renal, endocrine, neurologic, autoimmune, hepatic haematological (including pancytopenia, aplastic anaemia, or blood dyscrasia, etc.), metabolic (including diabetes mellitus), or pulmonary disease classed as significant by the Investigator.
   * History of any malignancy.
   * Systemic or local infection, such as the risk of sepsis and/or known active inflammation within 2 months before screening.
   * Severe infections requiring hospitalisation and/or the need for IV antibiotics, within 2 months before screening.
2. A sign of ongoing or chronic inflammation process defined as high blood concentration of C-reactive protein (CRP) (> 1.5 times the upper limit of normal [ULN]).
3. Subject has inadequate liver function as determined by following results:

   * Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 1.5 × ULN and
   * Total bilirubin > 1.5 × ULN.
4. Subject is considered to have a significant abnormal cardiac function in Investigator's discretion determined by the laboratory results.
5. Subject underwent surgical intervention or an operation within 4 weeks prior to the administration of the study drug (Day 1) or plans to undergo a surgical procedure during the study period.
6. Subject has active TB, latent TB (defined as a positive result for IGRA with no active lesion in examination of chest X-ray without any sign or symptom of TB), a history of TB, or had close contact with a person with active TB within 8 weeks prior to the administration of the study drug (Day 1). If the result of IGRA is indeterminate at screening, retest will be allowed only once during the screening period. If the repeated IGRA result is again indeterminate or positive, the subject will be excluded from the study. If the repeated IGRA result is negative, the subject may be included in the study.
7. Female subject is pregnant or lactating or planning to be pregnant or to breastfeed before, during, or within 5 months after the administration of the study drug (Day 1).
8. Male subject is planning to father a child or donate sperms within 5 months after the administration of the study drug (Day 1).
9. Subject has received a mAb or fusion protein within 9 months prior to randomization and/or there is a confirmed evidence or clinical suspicion of immunogenicity from previous exposure to a mAb or fusion protein, or subject is currently using a biologic (including but not limited to TNF-α blockers). Subjects with previous exposure to adalimumab are to be excluded.
10. Subject has received treatment with a biological or immunosuppressive agent (other than a mAb or fusion protein) within 3 months of screening.
11. Subject used prescription (excluding hormonal birth control), over the counter (OTC) drugs, dietary supplements, or herbal remedies that could affect the outcome of the study within 2 weeks prior to the administration of the study drug (Day 1).
12. Subject has undergone treatment with an investigational drug or participated in another clinical study for healthy subject or bioequivalence test within 90 days or 5 half-lives (whichever is longer) prior to the administration of the study drug (Day 1) or plan to do so during the study.
13. Subject received a live or live-attenuated vaccine within 4 weeks prior to the administration of the study drug (Day 1) or plan to do so until 6 months after Day 1.
14. Subject has donated or lost 450 mL or more of whole blood within 8 weeks, or donated blood components within 4 weeks prior to the administration of the study drug (Day 1).
15. Subject shows reasonable evidence of drug abuse (positive result for drug urine test and/or the opinion of the Investigator).
16. Subject has a history or presence of regular consumption exceeding an average weekly intake of 21 units of alcohol in recent 12 weeks prior to the screening visit. One unit is equivalent to a half-pint (285 mL) of beer/lager, one measure (25 mL) of spirits, or one small glass (125 mL) of wine. Subject is unwilling to avoid use of alcohol or alcohol containing foods, medications, or beverages within 24 hours prior to admission (Day -1), and each study visit until completion of the study.
17. Subject has smoked 10 or more cigarettes per day in the recent 12 weeks prior to the administration of the study drug (Day 1) and/or is unable to refrain from smoking up to 24 hours after the administration of the study drug.
18. In the opinion of the Investigator, the subject is not eligible for the study participation for any reason (including clinical laboratory results) or shows evidence of a condition (e.g., psychological, or emotional problem, any disorder or resultant therapy) that is likely to invalidate an informed consent or limit the ability of the subject to comply with the protocol requirements. Subject is unable to understand the protocol requirements, instructions, study-related restrictions, or the nature, scope, and possible consequences of the clinical study; or is unable to give written informed consent or to comply fully with the protocol.
19. Subject with confirmed COVID-19 infection by appropriate laboratory test screening and on admission.
20. Subject is vulnerable (e.g., employees of the study centre or any other individuals involved with the conduct of the study, or immediate family members of such individuals, persons kept in prison, or other institutionalised persons by law enforcement).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 324 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf) | Up to Day 71
  Primary endpoints were equivalence of PK between PBP1502 and reference drugs in terms of AUC0-inf. Blood samples for PK analysis were obtained pre-dose and at 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 192, 336, 504, 672, 1008, 1344, and 1680 hour post-dose.
Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-last) | Up to Day 71
  Primary endpoints were equivalence of PK between PBP1502 and reference drugs in terms of AUC0-last. Blood samples for PK analysis were obtained pre-dose and at 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 192, 336, 504, 672, 1008, 1344, and 1680 hour post-dose.
Maximum Serum Concentration (Cmax) | Up to Day 71
  Primary endpoints were equivalence of PK between PBP1502 and reference drugs in terms of Cmax. Blood samples for PK analysis were obtained pre-dose and at 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 192, 336, 504, 672, 1008, 1344, and 1680 hour post-dose.

SECONDARY OUTCOMES:
Time to the Maximum Serum Concentration (Tmax) | Up to Day 71
  The secondary objective was to evaluate the additional PK parameters of Tmax. Blood samples for PK analysis were obtained pre-dose and at 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 192, 336, 504, 672, 1008, 1344, and 1680 hour post-dose.
Terminal Elimination Half-life (t1/2) | Up to Day 71
  The secondary objective was to evaluate the additional PK parameters of t1/2. Blood samples for PK analysis were obtained pre-dose and at 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 192, 336, 504, 672, 1008, 1344, and 1680 hour post-dose.
Adverse events | Up to Day 71
  Adverse events will be coded using MedDRA and grouped by system organ class and preferred term and summarised, by treatment group at the time of onset of the AE. The summary tables will present the number and percentage of total subjects and number of events, by system organ class and by preferred term. Injection related reactions will be listed and summarised by reaction using frequency counts and percentage, by treatment group.
Anti Drug Antibodies (ADAs) | Up to Day 71
  Formation of Anti Drug Antibody will be measured through a validated assay.
Neutralizing Antibodies (NAbs) | Up to Day 71
  Formation of neutralizing antibodies measured through a validated system

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Fase I. U. Autonoma de Madrid (Clinical Trials Unit, UAM) C/ Arzobispo Morcillo 4, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No